CLINICAL TRIAL: NCT00726362
Title: To Explore the Treatment Effect of Various Commercially Available Statins on Patients With Hyperlipidemia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: William Huang/Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CTW-CRE-2007/1
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Hyperlipidemias
Keywords: Statin; LDL-C
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with hyperlipidemia newly initiating a statin; or switched from current therapy to a statin, or require dosage adjustment for statin

SUMMARY:
The primary objective is to survey the efficacy of various commercially available statins (a class of lipid-lowering agents, for example, rosuvastatin, atorvastatin, simvastatin, lovastatin, pravastatin and fluvastatin) under local clinical practice in treating patients with hyperlipidemia. Surveillance data (Lipid Profile) will be collected during course of usual clinical practice or captured upon its availability.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with hyperlipidemia
* Patients who are just starting a statin treatment, who need to switch from current therapy to a statin medication, or who are receiving dosage adjustment of statin as judged by the physicians
* Patients who are willing to participate in this study and who sign an informed consent form

Exclusion Criteria:

* Pregnancy or breast feeding
* Patient are illiterate or unable to fill the questionnaire for any reason
* Patients with contraindications to the use of certain statins as needed prescribed by physicians (as per commercially available statins package insert) including the use of rosuvastatin.
* Any clinical condition which, in the opinion of the attending physician, would not allow safe administration of the study medications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: based on regular practice and judged by physicians, patients with hyperlipidemia who need to start prescribed with a statin; or to switch from current therapy to a statin, or require dosage adjustment for statin
Sampling Method: Probability Sample
Enrollment: 3270 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Changes on LDL-C, HDL-C, TG, TC | 3~6 months

SECONDARY OUTCOMES:
ratio for treatment-to-goal | 3~6 months
drug compliance | 3~6 months
correlation between patient's insight and therapeutic outcome | 3~6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ter Lai, MD, Principal Investigator — Kaohsiung Medical University
Locations (8):
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Douliu
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Pingtung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei